CLINICAL TRIAL: NCT00874146
Title: Retrospective Study of the Level of HER2-neu Gene Amplification as Predictive Factor of Response in Patients With HER2-positive Advanced Breast Cancer Treated With Trastuzumab Containing Regimens.
Brief Title: Level of HER2-neu Gene Amplification an Response to Trastuzumab
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Armando Santoro, MD, Istituto Clinico Humanitas
Other Study IDs: ONC/OSS-03-2008
Record Dates: First submitted 2009-03-26; First posted 2009-04-02 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-09

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — In Situ Hybridization, Fluorescence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FISH test performed on paraffine embedded tumor sections.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: HER2-positive advanced breast cancer
  Interventions: Genetic: Fluorescent in-situ hybridization (FISH)

INTERVENTIONS:
Genetic: Fluorescent in-situ hybridization (FISH) — Dual color FISH test to assess ratio of HER2/neu amplification

SUMMARY:
Primary objective of the study is to evaluate the correlation between level of HER2-neu gene amplification evalued by dual-color Fluorescent in-situ hybridization (FISH) test and time to progression (TTP) in patients with HER2-positive advanced breast cancer treated with trastuzumab-containing regimens.

ELIGIBILITY:
Inclusion Criteria:

* HER2-positive breast cancer Trastuzumab-containing regimen delivered for advanced disease Tumor sample available at Pathology Archive

Exclusion Criteria:

* HER2-negative advanced breast cancer Pretreatment with trastuzumab

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2-positive advanced breast cancer treated with trastuzumab-containing regimen.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Association of tumor cytogenetic paremeters with TTP and OS. | one year

SECONDARY OUTCOMES:
Association of cytogenetic parameters evalued by FISH test and patients' characteristics. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinco Humanitas, Rozzano, Milan, Italy